CLINICAL TRIAL: NCT06657326
Title: Evaluation of the Efficacy (QCA) and Safety of the BioFreedom™ Ultra Drug Coated Stent in Patients With High Bleeding Risk and Coronary Artery Disease Undergoing Percutaneous Coronary Intervention
Brief Title: LEADERS FREE IV (RCT): BioFreedom™ Ultra vs BioFreedom™ in HBR Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-AP-01
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Disease; Chronic Stable Angina; Unstable Angina; Silent Ischemia; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable; Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Patient will be randomized to one of the treatment arms to receive either the BioFreedom™ Ultra DCS or BioFreedom™ DCS
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioFreedom™ Ultra DCS (Experimental): Coronary artery disease patients with high-bleeding risk (HBR) will receive the BioFreedom™ Ultra stent if randomized to this arm (1:1 ratio)
  Interventions: Device: BioFreedom™ Ultra cobalt-chromium Biolimus A9™-coated stent
- BioFreedom™ DCS (Active Comparator): Coronary artery disease patients with high-bleeding risk (HBR) will receive the BioFreedom™ stent if randomized to this arm (1:1 ratio)
  Interventions: Device: BioFreedom™ stainless steel Biolimus A9™-coated stent

INTERVENTIONS:
Device: BioFreedom™ Ultra cobalt-chromium Biolimus A9™-coated stent — Stent implantation
  Arms: BioFreedom™ Ultra DCS
Device: BioFreedom™ stainless steel Biolimus A9™-coated stent — Stent implantation
  Arms: BioFreedom™ DCS

SUMMARY:
This study aims to demonstrate that the BioFreedom™ Ultra Drug Coated Stent (DCS) is non-inferior to the BioFreedom™ DCS, with respect to in-stent late lumen loss, and that it has safety characteristics similar to the BioFreedom™ DCS.

DETAILED DESCRIPTION:
The LEADERS FREE IV trial is conducted to evaluate of the efficacy (QCA) and safety of the BioFreedom™ Ultra Drug Coated Stent in patients with High Bleeding Risk (HBR) and coronary artery disease undergoing Percutaneous Coronary Intervention.

It is a prospective, multi-center, single blind (to patient), randomized, comparator trial, designed to randomize 444 HBR patients at approximately up to 7 centers in Malaysia.

The primary objective is to confirm non-inferiority of the BioFreedom™ Ultra stent compared to BioFreedom™ DCS as measured by the difference in angiographically measured late lumen loss at 9 months, and the main secondary objective is to assess safety as measured by TLF and ST. 444 patients will be randomized 1:1 to either stent, allowing for a direct comparison, and will be followed up to 5 years to measure for late TLF and ST events.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at high bleeding risk (HBR) with an indication for PCI who can tolerate at least one month of DAPT. This includes patients with stable angina, silent ischemia, acute coronary syndromes (ACS) (STEMI and NSTEMI), de novo lesions in native arteries with diameter stenosis >70% by visual estimation and evidence of ischemia in the territory of the target vessel(s).
2. Patients meet ARC-HBR definition i.e at least 1 major or 2 minor criteria.

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Age <18 years old
3. Patients lacking capacity (i.e. patients suffering from dementia and others) to provide informed consent
4. Patients expected not to comply with 1 month DAPT
5. Active bleeding at the time of inclusion
6. Procedure requires the use of non-study stents, or alternative therapeutic options not followed by stent implantation (angioplasty only, atherectomy only)
7. Number of target lesions >2
8. Patient requires a stent of diameter <2.25mm
9. Patient requires a stent of diameter >4.0mm
10. Isolated ostial lesions within 3 mm of the origin of LAD or LCx (left main lesions involving the ostia of the LAD and/or LCx are eligible)
11. Patient has known left ventricular ejection fraction (LVEF) <30% (LVEF may be obtained at the time of the index procedure if the value is unknown and the investigator believes it is necessary)
12. Patient with chronic total occlusion(s) as target lesion(s)
13. Severe calcification that might prevent sufficient expansion of the DES, unless pre-treated with a plaque modification device such as cutting balloon, scoring balloon or intravascular lithotripsy.

    Note: Use of rotational or orbital atherectomy is also permitted.
14. Cardiogenic shock
15. Compliance with long-term single anti-platelet therapy unlikely
16. Known hypersensitivity or contraindication to aspirin, clopidogrel (or to any other P2Y12 inhibitor if applicable), cobalt chromium, stainless steel, zinc, Biolimus A9™ or a sensitivity to contrast media, which cannot be adequately pre-medicated
17. Any PCI during the previous 12 months
18. Participation in another clinical study (12 months after index procedure)
19. Patients with a life expectancy of <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
In-stent late lumen loss (LLL) at 9 months | 9 months
  In-stent late lumen loss (LLL) assessed by quantitative coronary angiography (QCA) at 9 months

SECONDARY OUTCOMES:
All clinical events at protocol defined timepoints | 1,6,9,12 months, 2 ,3, 4, 5 years
  * Cardiovascular Death
  * Myocardial infarction (according to the Fourth Universal Definition)
  * TLF (defined as cardiovascular death, target vessel related MI and clinically driven (cd) target lesion revascularization (TLR))
  * All-cause mortality
  * Clinically driven TVR
  * Stent Thrombosis, per ARC-2 definition of definite/probable
  * Device success
  * Procedure success
  * Lesion success
  * Bleeding per BARC criteria
    * BARC 3 to 5
    * All BARC
    * By vascular access site (Femoral/Radial)

CONTACTS AND LOCATIONS:
Overall Officials: Kamaraj a/l Selvaraj, Dr., Principal Investigator — Hospital Serdang
Locations (6):
- Malaysia (6):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Queen Elizabeth II, Kota Kinabalu, Sabah
  - Pusat Jantung Hospital Umum Sarawak, Kota Kinabalu, Sarawak
  - Hospital Serdang, Kajang, Selangor

IPD SHARING:
Plan to Share IPD: No
Data relating to the study might be made available to third parties provided the data are treated confidential and that the patient's privacy is guaranteed.